CLINICAL TRIAL: NCT03629197
Title: A Clinician Training Intervention to Improve Pain-related Communication, Pain Management and Opioid Prescribing in Primary Care
Brief Title: Improving Communication About Pain and Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 970014; 5K23DA043052 (NIH); A18-0560 (Other: UC Davis)
Record Dates: First submitted 2018-07-31; First posted 2018-08-14 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Pain, Chronic; Communication Research; Opioid Use
Keywords: primary care; chronic pain; patient-physician communication; opioid analgesics; standardized patients
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Physicians will be randomized to receive the intervention versus control; patients will be recruited to see study physicians; patients will not be randomized.
Masking Description: Physicians will be randomized after physician recruitment is complete. This ensures that arm assignment does not impact physicians' decision to participate. Arm assignment will be done using a random number generator. Due to the nature of the intervention, blinding participants (physicians) is not feasible. However, patients will not be aware of their physician's arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication skills training (Experimental): Intervention clinicians will receive 2 standardized patient visits. The first visit will consist of an 8 minute video on the development of 5 key communication skills, a 10-12 minute role-play session to practice using these skills, and 8-10 minutes of constructive feedback. The 2nd visit will include only the role-play and feedback components. Clinicians will also get a printed pocket card and pamphlet explaining the targeted communication skills in more detail.
  Interventions: Behavioral: Communication skills training
- Control (Active Comparator): Control clinicians will receive a written summary of the 2016 CDC opioid prescribing guidelines, which include recommendations for best practices for use of opioids to treat chronic non-cancer pain. CDC guidelines will serve as an attention control.
  Interventions: Other: Attention control

INTERVENTIONS:
Behavioral: Communication skills training — Intervention components include an 8-10 minute instructional video, a pocket card and pamphlet, and 2 standardized patient visits with role-play and feedback by the standardized patient
  Arms: Communication skills training
Other: Attention control — Physician will review materials based on CDC opioid prescribing guidelines.
  Arms: Control

SUMMARY:
The overall goal of this protocol is to pilot test a clinician training intervention that uses standardized patients (trained actors playing patient roles) as instructors who impart communication skills to primary care clinicians. This project will conduct a pilot clinical trial of the intervention developed by the primary investigator in order to evaluate intervention feasibility and generate data to plan a subsequent fully-powered, multisite trial. Primary care clinicians will be randomized to receive either the intervention or control; 48 patients (2 per clinician) will then be recorded during clinic visits with study clinicians and will provide data on post-visit perceptions and health outcomes. Study hypotheses are that visits with clinicians who receive the intervention (versus control) will be associated with more frequent use of targeted communication skills, lower probability of high-risk opioid prescribing, higher patient-reported agreement with treatment plan, and lower pain interference 2 months later.

DETAILED DESCRIPTION:
The only intervention in the randomized controlled trial (RCT) will be clinician education. This RCT will not directly manipulate or influence patient care. Therefore, this study is minimal risk. The only foreseeable patient risks relate to data confidentiality and privacy.

The investigators will recruit approximately 48 primary care clinicians for the pilot RCT. The study goal is to enroll 24 residents and 48 patients (2 patient visits per resident). However, based on previous experience with similar recruitment methods in these clinics, only about 50% of enrolled clinicians will ultimately have visits with study patients. Thus, it will be necessary to over-enroll clinicians because the investigators expect a large proportion of residents will have to be dropped from study due to not seeing any study patients. After enrollment, clinicians will complete a brief questionnaire including demographics and self efficacy regarding communicating with patients about chronic pain and opioids.

Randomization assignment will take place after all clinicians have provided informed consent and enrolled, to prevent randomization status from influencing enrollment decisions. Randomization assignment will be done by study personnel after all clinicians have been recruited. Randomization is at the clinician level. Because of the nature of the intervention, it is not possible to blind subjects or investigators to randomization assignment. However, patients will be unaware of clinicians' randomization assignment.

Intervention clinicians will complete 2 standardized patient visits during regular clinic time. The first visit will include viewing an 8-10 minute video summarizing the key communication skills, a 10-12 minute roll-play session to practice using these skills, and 8-10 minutes of constructive feedback. The second video will have only roll-play and feedback. Control clinicians will receive a written summary of the 2016 Centers for Disease Control and Prevention (CDC) opioid prescribing guidelines which include recommendations for best practices for use of opioids to treat chronic non-cancer pain. To the extent possible, the investigators will use CDC-produced materials for the control group. CDC guidelines will serve as an attention control. Intervention clinicians will complete a brief questionnaire evaluating the intervention. Some time later, enrolled clinicians will see 2 patients who've been screened and enrolled by the research team and who've agreed to allow a previously scheduled visit with pcp to be audio recorded. Data will include the audio recording transcripts, a pre-visit and post-visit patient questionnaire and a clinician post-visit questionnaire.

2 months after each patient's visit, a research assistant will call patients and obtain 2-month follow up data (e.g. Brief Pain Inventory).

ELIGIBILITY:
Inclusion Criteria:

Internal Medicine or Family Medicine residents at UC Davis:

* completed ≥1 year of training
* see primary care patients in the Ambulatory Care Center (ACC) building. Clinicians will be recruited through clinic huddles, emails, and presentations at meetings.

UC Davis Patients:

* 18-80 years old
* taking opioids (≥1 opioid dose per day) prescribed by their primary care physician for >90 days to treat chronic musculoskeletal pain
* have an appointment scheduled with a participating clinician at which they report they are likely to discuss pain management

Exclusion Criteria:

* active cancer
* hospice
* do not speak English
* prisoners
* pregnant women
* unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Clinician use of targeted communication skills | Over a 3-9 month period (depending on how soon after the intervention clinicians' appointments with patient participants can be scheduled).
  Compare frequency of use of targeted communication skills for residents in the Intervention vs Control arm (using coding of recorded visits to assess skill use)
Compare efficacy of Control vs Intervention by measuring changes in the way pain interfered with patients lives using the Brief Pain Inventory - Pain Interference subscale survey | 8 weeks
  Brief Pain Inventory (BPI) Pain Interference subscale consists of 7 categories relating to how pain interferes with patients lives. Patients are asked to rate their pain on a zero (Does Not Interfere) to 10 (Completely Interferes) scale. The 7 categories are: 1. General Activity, 2. Mood, 3. Walking Ability, 4. Work, 5. Relationships, 6. Sleep, 7. Enjoyment of life. Results are averaged to give an overall interference rating

SECONDARY OUTCOMES:
Compare efficacy of Control vs Intervention by measuring changes in the severity of patients pain using the Brief Pain Inventory - (Short Form) Pain Severity subscale which measures the severity of the patient's pain. | 8 weeks
  Brief Pain Inventory (BPI) Short Form -- Pain Severity subscale has 4 survey questions / categories, asking patients to rate the severity of their pain on a 0-10 scale (with 0 being No Pain and 10 being Worst Possible Pain). The 4 Categories are, A. At it's worst in the last 24 hours, B. At it's best in the last 24 hours, C. Pain on average, D. Pain right now. Results are averaged to give an overall score.
Difficult Doctor-Patient Relationship Questionnaire | Over a 3-9 month period (depending on how soon after the intervention clinicians' appointments with patient participants can be scheduled).
  Comparison of difficult doctor-patient encounter scale for Intervention vs Control physicians. Difficult doctor-patient relationship scale has 10 items scored from 1-6 . The overall scale range is 10-60, with higher values indicating more difficult visits.
Patient experience score | 8 weeks
  Difference in patient experience for patients who saw Intervention vs Control physicians (measured by post-visit patient agreement with treatment plan, patient trust, and patient assessment of clinician communication skills). Patient experience will be a "standardized average" of 3 different scales:
  1. Patient assessment of physician communication skills is a subscale of the CAHPS (Consumer Assessment of Health Plan Survey) Adult Visit Survey. Range is 0-12, with higher indicating better communication skills.
  2. Patient agreement with treatment plan scale. Range is 3-21, with higher being greater agreement).
  3. Brief Wake Forest Patient Trust in Physician Scale. Range is 5-25, with higher being greater trust.
Physicians' overall appraisal of the standardized patient Intervention | 1-3 months
  Physician reported assessment of intervention. Investigators will ask for physicians' evaluation of the feasibility, acceptability, and utility of the intervention. Investigators will offer 10 value statements about the intervention. Physicians will select 1 from the following choices: strongly agree, agree, neutral, disagree, strongly disagree. Results will be averaged to give an overall score; higher values indicate more positive appraisal.
Change in physician communication self efficacy | Over 3-9 month period (depending on how soon after the intervention clinicians' appointments with patient participants can be scheduled).
  Change in physician self efficacy for communication skills for Intervention vs Control physicians. These questions ask about physicians' confidence related to managing chronic non-cancer pain in primary care. Physicians will be asked to rate how strongly they agree or disagree with each statement. Higher values indicate greater self efficacy. Baseline and post-visit ratings of self efficacy will be computed, and we will measure change in self efficacy (post-visit self efficacy minus baseline self efficacy) for Control vs Intervention physicians.

OTHER OUTCOMES:
High-risk opioid prescribing | Over 3-9 month period (depending on how soon after the intervention clinicians' appointments with patient participants can be scheduled).
  Prevalence of high-risk opioid prescribing as measured by chart review

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G Henry, MD, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis Family Medicine Clinic, Sacramento, California
  - University of California Davis Internal Medicine Clinic, Sacramento, California

IPD SHARING:
Plan to Share IPD: No